CLINICAL TRIAL: NCT03408951
Title: Surface ECG Signal Recording for the Implantable Subcutaneous String Defibrillator (ISSD) Detection Algorithm Performance Assessment
Status: Completed | Type: Observational
Sponsor: NewPace Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NPC03
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2018-01

CONDITIONS: Tachyarrhythmia; Arrhythmias, Cardiac
MeSH Terms: conditions — Tachycardia; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventions (recording): Patients requiring Intracardiac defibrillator (ICD) implantation or Defibrillation Test (DFT) or Electrophysiology (EP) study with high probability of supra ventricular tachyarrhythmia.
  Interventions: Other: Recording

INTERVENTIONS:
Other: Recording — The patient cutaneous ECG is recorded, to later be comparatively analysed by an expert and by the ISSD detection algorithm

SUMMARY:
Recorded cutaneous ECG containing arrhythmia events are separately analysed by an expert Electrophysiologist and the ISSD detection algorithm, to allow assessment of the correct detection of tachyarrhythmia events and discrimination of supra-ventricular arrhythmia of the algorithm,m compared to the expert.

DETAILED DESCRIPTION:
cutaneous ECG electrodes positioned near the sternum and on the midaxillary line, at the approximate positions of the ISSD sense electrodes, are used to record patients undergoing Defibrillation Threshold (DFT) studies or Electrophysiology (EP) studies of different types. Two separate copies of the recordings undergo parallel and separate analysis: one is sent to an expert Electrophysiologist for determination and classification of arrhythmia events of at least 5 seconds and at least 170 beats per minute. the other is fed to the ISSD detection algorithm, with a low cutoff rate of 170 beats per minute. the results are compared to establish the accuracy of the detection algorithm and the rate of false detection / classification of arrhythmia events.

ELIGIBILITY:
Inclusion Criteria:

* candidate for ICD implantation
* candidate for an ICD DFT study
* candidate for an EP study

Exclusion Criteria:

* age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high chance of having a cardiac tachyarrhythmia
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
ISSD algorithm detection rates | through study completion, expected at 15 months
  Calculation of the ISSD algorithm detection and classification rates, compared to an EP expert analysis of the ECG traces

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H Levine, M.D, Principal Investigator — St Francis Hospital Heart Center; David Hoch, M.D, Principal Investigator — St Francis Hospital Heart Center
Locations (1):
- St Francis Hospital Heart Center, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No